CLINICAL TRIAL: NCT02626962
Title: Phase II Multicenter, Non Randomized, Open Label Trial of Nivolumab in Combination With Ipilimumab in Subjects With Previously Untreated Metastatic Uveal Melanoma
Brief Title: Trial of Nivolumab in Combination With Ipilimumab in Subjects With Previously Untreated Metastatic Uveal Melanoma
Acronym: GEM1402
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-1402; 2015-004429-15 (EudraCT Number)
Record Dates: First submitted 2015-12-01; First posted 2015-12-10 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Uveal Melanoma
Keywords: melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab and Ipilimumab (Experimental): Nivolumab and Ipilimumab every 3 weeks for a total of four doses (Cycles 1 and 2) followed by Nivolumab every 2 weeks
  Interventions: Drug: ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: ipilimumab — Ipilimumab every 3 weeks for a total of four doses (Cycles 1 and 2)
  Other Names: Yervoy
Drug: Nivolumab — Nivolumab every 3 weeks for a total of four doses (Cycles 1 and 2) followed by Nivolumab every 2 weeks
  Other Names: Opdivo

SUMMARY:
This is a Phase 2, single-arm study of nivolumab combined with ipilimumab in subjects with previously untreated, unresectable or metastatic uveal melanoma. Previous studies with immunotherapy have shown promising results and this synergistic combination was very effective in other tumors. This study will allow for further characterization of the safety and clinical activity of nivolumab combined with ipilimumab in subjects with uveal melanoma.

DETAILED DESCRIPTION:
Uveal melanoma is a rare disease, accounting for 0.1% of all cancer deaths. This disease arises from melanocytes of the uveal tract and is the most common primary intraocular tumor in adults, with an incidence estimated at 0.6 per 100,000 persons/year in the Western population and seems to have remained stable over time.

Metastases in uveal melanoma appear in 6.5%-35% of the patients during the first decade. The clinical and metastatic behavior differs from cutaneous melanoma because of its initially purely hematogenous dissemination and its tendency to metastasize to the liver. Furthermore, the liver is almost a "sentinel lymph node" for uveal melanoma, because it is affected in 95% of patients and it is the sole site of metastasis in most cases. This specific ocular-hepatic tropism remains unexplained. When liver metastases develop, the prognosis is poor and life expectancy is reduced to less than 6 months in the absence of treatment. Only few prognostic factors for survival have been identified. Age, short time interval to metastases development, and tumor burden in the liver have shown a negative impact on survival, whereas patients diagnosed at regular follow-up survive significantly longer, probably due to the earlier diagnosis. Several loco-regional treatment options can be considered if metastases are confined to the liver, including partial hepatic resection or radiofrequency ablation. Curative resection is possible in only a small fraction of patients due to the number, location or size of the metastases.

Systemic chemotherapy is usually unsuccessful in metastatic uveal melanoma and results were recently reviewed showing an Overall Response Rate of 4,6 %with 95% CI 3.3-6.3%. There is no proof that conventional chemotherapy prolongs survival with most studies reporting OS between 5 and 12 months. Most therapies are derived from the experience extrapolated from cutaneous melanoma. Only few chemotherapeutic regimens have been studied in phase II trials such as bleomycin /vincristine/ lomustine /dacarbazine (BOLD), fotemustine,9-nitrocamptothecin, temozolomide, bendamustine, gemcitabine/treosulfan, cisplatin/gemcitabine/treosulfan, and dacarbazine/treosulfan with poor results that range from 0 to 15% response rate and less than 12 months overall survival with first line therapy. A phase III trial randomizing patients to chemotherapy or Best Suportive Care (BSC) is not expected to be performed because of difficulty in recruiting due to the low incidence of disease.

In the other hand, the best understanding of the biology of cancer disease has allowed us to identify pathways that are important in mechanisms of proliferation, survival or dissemination. Recently Guanine Nucleotide-Binding Protein G (GNAQ) gene oncogenic mutation has been identified in close to 50% of primary uveal melanomas. The emergence of newer agents that target this or other pathways (such as selumetinib, sunitinib, imatinib, vorinostat, antiangiogenics) have resulted in multiple small studies that up to date have failed to show a clear superiority against chemotherapy. To summarize, patients with metastatic uveal melanoma should be included in clinical trials evaluating other options with newer agents with potentially less toxicity and greater efficacy than conventional chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be provided;
2. Patients must have a histological diagnosis of uveal melanoma;
3. Progressive metastatic disease at baseline. Progressive disease is defined as new or progressive lesions on cross-sectional imaging;
4. Age>18 years;
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 1;
6. Measurable disease by CT or MRI per RECIST 1.1 criteria;

Exclusion Criteria:

1. Prior systemic treatment for metastatic uveal melanoma.
2. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of cervix or breast, or incidental prostate cancer.
3. Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis). Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
4. Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of nivolumab and ipilimumab hazardous or obscure the interpretation of Advers Events (AEs), such as a condition associated with frequent diarrhea.
5. Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of nivolumab and ipilimumab).
6. A history of prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
7. Concomitant therapy with any of the following: Interleukin (IL) -2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids, defined as >10mg daily prednisone equivalents. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
8. Active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 8 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
9. Women of childbearing potential (WOCBP) as defined below, who:

   * are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 8 weeks after cessation of study drug, or
   * have a positive pregnancy test at baseline, or
   * are pregnant or breastfeeding.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Overall Survival at 12 months | 12 months after treatment start
  Percentage of patients alive at 1-year from first dose of treatment.

SECONDARY OUTCOMES:
Overall survival at 24 months. | 24 months
  Percentage of patients alive at 2-years from first dose of treatment.
Progression Free Survival (PFS) | 3 months
  Percentage of patients without progression of disease at month 3, according RECIST 1.1 criteria.
Global PFS according to RECIST 1.1 criteria. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Percentage of patients without progression of disease at month throughout follow-up, according RECIST 1.1 criteria.
Objective Response Rate (ORR) | 12 months
  Respose to treatment according to RECIST 1.1 criteria
Disease Control Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Percentage of patients with disease control
Duration of response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Length of time between date of evidenced response and progression of disease or death

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Piulats, MD, Study Chair — ICO Hospitalet
Locations (10):
- Spain (10):
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - ICO Hospitalet, L'Hospitalet de Llobregat
  - H. Insular de Canarias, Las Palmas de Gran Canaria
  - Hospital La Paz, Madrid
  - H. U. Virgen de la Victoria, Málaga
  - Clínica Universidad de Navarra, Pamplona
  - H. U. Clínico de Santiago, Santiago
  - H.U. Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia
  - H. C. U. de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Piulats JM, Espinosa E, de la Cruz Merino L, Varela M, Alonso Carrion L, Martin-Algarra S, Lopez Castro R, Curiel T, Rodriguez-Abreu D, Redrado M, Goma M, Rullan AJ, Calvo Gonzalez A, Berrocal-Jaime A. Nivolumab Plus Ipilimumab for Treatment-Naive Metastatic Uveal Melanoma: An Open-Label, Multicenter, Phase II Trial by the Spanish Multidisciplinary Melanoma Group (GEM-1402). J Clin Oncol. 2021 Feb 20;39(6):586-598. doi: 10.1200/JCO.20.00550. Epub 2021 Jan 8. PMID 33417511